CLINICAL TRIAL: NCT01349829
Title: A Phase IV Open, Randomized, Controlled Study to Evaluate the Safety and Immunogenicity of a Pediatric Presentation (0.25 ml) of the Virosomal Hepatitis A Virus (HAV) Vaccine HAVpur in Healthy Young Children Aged Between and Including 18 Months to 47 Months, Using a 0/6 Month Immunization Schedule
Brief Title: A Study to Evaluate the Safety and Immunogenicity of the Hepatitis A Virus Vaccine HAVpur in Healthy Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPA-V-A008
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis A
Keywords: Hepatitis A; Vaccination; Immunity
MeSH Terms: conditions — Hepatitis A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAVpur (Experimental)
  Interventions: Biological: HAVpur Junior
- Havrix (Active Comparator)
  Interventions: Biological: Havrix 720 Junior

INTERVENTIONS:
Biological: HAVpur Junior — ≥12 International Units (IU) hepatitis A antigen coupled to virosomes, intramuscularly (i.m.), anterolateral thigh (M. vastus lateralis) or deltoid (M. deltoideus)
  Vaccination schedule: single doses at 0 and 6 months
  Arms: HAVpur
Biological: Havrix 720 Junior — ≥720 ELISA Units (EU) hepatitis A antigen adsorbed to aluminium hydroxide, intramuscularly (i.m.), anterolateral thigh (M. vastus lateralis) or deltoid (M. deltoideus)
  Vaccination schedule: single doses at 0 and 6 months
  Arms: Havrix

SUMMARY:
This is a study to test whether vaccination with HAVpur Junior against hepatitis A provides protection that is non-inferior to the protection afforded by vaccination with Havrix 720 Junior.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between (and including) 18 months to 47 months of age.
* Written informed consent obtained from the parent/legal guardian of the subject.
* Free of obvious health problems as established by medical history and/or clinical examination before entering the study

Exclusion Criteria:

* Seropositive for anti-HAV antibodies (>=10 mIU/ml).
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and safety follow-up.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose (for corticosteroids, such as prednisone, or equivalent, >=0.5 mg/kg/day.
* Inhaled and local steroids are allowed.)
* Planned administration/ administration of a measles containing vaccine within 4 weeks prior to and after the first or booster dose of study vaccine.
* Previous vaccination against hepatitis A.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment

Ages: 18 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daljit Singh, MD, Principal Investigator — Dayanad Medical College and Hospital; Tejinder Singh, MD, Principal Investigator — Christian Medical College and Hospital; Hemant Jain, MD, Principal Investigator — Medical College and Chacha Nehru Bal Chikitsalay; Vardana Kumavat, MD, Principal Investigator — Rajiv Ghandi Medical College
Locations (3):
- India (3):
  - Medical College and Chacha Nehru Bal Chikitsalay, Indore, Madhya Pradesh
  - Rajiv Ghandi Medical College, Thane, Maharashtra
  - Christian Medical College and Hospital, Ludhiana, Punjab

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 25 March 2010 to 18 April 2011; outpatient study
Period: Overall Study
Arm/Group | HAVpur | Havrix
Started | 126 | 125
Completed | 117 | 102
Not Completed | 9 | 23
Not completed — Lost to Follow-up | 4 | 8
Not completed — Consent withdrawal | 3 | 8
Not completed — Migrated/moved | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HAVpur | Havrix | Total
Number analyzed (Participants) | 126 | 125 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 126 | 125 | 251
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: months] | 27.6 (8.45) | 27.9 (8.23) | 27.8 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 68 | 127
  Male | 67 | 57 | 124

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection at Month 1
Description: Proportion of subjects seroprotected (seroprotection defined as anti-HAV antibody concentration >=10 mIU/ml)
Time Frame: Month 1
Population: Results are for the ATP population included all randomized subjects who received the first vaccination and had negative anti-HAV antibody concentration at screening, and who had no major protocol violations and whose serum sample after the first vaccination was available for measurement of immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 122 | 117
percentage of participants | 95.9 [90.7 to 98.7] | 96.6 [91.5 to 99.1]

2. Secondary Outcome: Seroprotection at Month 6
Description: Proportion of subjects seroprotected (>=10 mIU/ml)
Time Frame: Month 6
Population: Results are for the ATP population included all randomized subjects who received the first vaccination and had negative anti-HAV antibody concentrations at screening, no major protocol violations and whose serum sample was available for measurement of immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 115 | 105
percentage of participants | 98.3 [93.9 to 99.8] | 99.0 [94.8 to 100]

3. Secondary Outcome: Seroprotection at Month 7
Description: Proportion of subjects seroprotected (>=10 mIU/ml)
Time Frame: Month 7
Population: Results are for the ATP population included all randomized subjects who received the first and second vaccination and had negative anti-HAV antibody concentrations at baseline, no major protocol violations and whose serum sample after the second vaccination was available for measurement of immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 112 | 94
percentage of participants | 100 [96.8 to 100] | 100 [96.2 to 100]

4. Secondary Outcome: Geometric Mean Concentrations (GMCs)
Description: GMCs of anti-HAV antibodies will be measured from blood samples
Time Frame: Month 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 122 | 117
mIU/mL | 51.5 [41.5 to 64.0] | 53.3 [42.8 to 66.5]

5. Secondary Outcome: Geometric Mean Concentrations (GMCs)
Description: GMCs of anti-HAV antibodies will be measured from blood samples
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 115 | 105
mIU/mL | 96.0 [71.8 to 128.4] | 113.0 [83.7 to 152.5]

6. Secondary Outcome: Geometric Mean Concentrations (GMCs)
Description: GMCs of anti-HAV antibodies will be measured from blood samples
Time Frame: Month 7
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HAVpur | Havrix
Number analyzed (Participants) | 112 | 94
mIU/mL | 1712.4 [1377.1 to 2129.3] | 2226.4 [1758.4 to 2819.1]

ADVERSE EVENTS:
Arm/Group | HAVpur - First Vaccination | Havrix - First Vaccination | HAVPur - Second Vaccination | Havrix - Second Vaccination
Serious Adverse Events (participants affected / at risk) | 0/126 | 1/125 | 1/118 | 0/108
Other Adverse Events (participants affected / at risk) | 24/126 | 24/125 | 4/118 | 6/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAVpur - First Vaccination (N=126) | Havrix - First Vaccination (N=125) | HAVPur - Second Vaccination (N=118) | Havrix - Second Vaccination (N=108)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAVpur - First Vaccination (N=126) | Havrix - First Vaccination (N=125) | HAVPur - Second Vaccination (N=118) | Havrix - Second Vaccination (N=108)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (solicited) (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (solicited) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (solicited) (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (solicited) (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (unsolicited) (General disorders) | 5 (5) | 5 (6) | 1 (1) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No